CLINICAL TRIAL: NCT01099943
Title: Reducing Inappropriate Antibiotic Prescribing by Primary Care Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-1022; HHSA290200710008
Record Dates: First submitted 2009-11-03; First posted 2010-04-08 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Increased Drug Resistance; Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Education, Decision Support Tools (Experimental): Clinic sites randomized to the intervention group will participate in an educational intervention comprised of lectures on antimicrobial resistance and implement decision support tools to guide primary care providers in appropriate antibiotic prescribing for common infectious conditions.
  Interventions: Other: Intervention: Education, Decision Support Tools
- No education, no implemented decision support tools (No Intervention): Clinics randomized to the control will not participate in the education intervention and implementation of decision support tools.

INTERVENTIONS:
Other: Intervention: Education, Decision Support Tools — Clinic sites randomized to the intervention group will participate in an educational intervention comprised of lectures on antimicrobial resistance and implement decision support tools to guide primary care providers in appropriate antibiotic prescribing for common infectious conditions.
  Arms: Intervention: Education, Decision Support Tools

SUMMARY:
Hypotheses and Specific Aims:

The continued emergence of antibiotic-resistance in the outpatient setting underlines the need to responsibly manage antimicrobial prescribing. It is in this context that we seek to test an effective strategy for reducing the inappropriate use of antibiotics in primary care office practices. Our overall objective is to identify an effective and efficient strategy for decreasing the contribution of primary care clinicians to the emergence of antimicrobial-resistant bacteria in the community and to disseminate widely those strategies found to be effective and sustainable.

We hypothesize that implementation of a clinician decision support system, with an active education component, will reduce the inappropriate use of antibiotics in primary care office practices. Our hypothesis is based on the premise that most inappropriate prescribing is the result of multiple factors that include difficulty in distinguishing a benign, self-limited viral infection from a more serious bacterial infection; overdiagnosis of a bacterial infection in cases where there is clinical uncertainty as to the true nature of the illness; and constraints on the time available for clinicians to explain to patients the nature of the illness and the reasons an antibiotic is not indicated.

The focus of this proposal will be to compare the impact of clinical decision support and active education to no intervention for enhancing the appropriate use of antimicrobials for common outpatient infections. In this randomized control trial, primary care providers participating in the intervention arm will receive active education coupled with the implementation of a clinical decision support tool, while providers in the control arm will have no intervention. At the end of the study, providers in the control arm will receive a thorough analysis of their antibiotic prescribing patterns and suggested opportunities for improvement, as well as access to the intervention tools once the study has ended.

Our interdisciplinary team will integrate novel methods in implementation science with clinical and laboratory expertise in infectious diseases, antimicrobial stewardship, primary care, information technology, performance improvement, health services research, and biostatistics. The Specific Aims are constructed to validate our hypothesis in the primary care setting by demonstrating two results of our intervention strategy:

1. Reduced use of antibiotics to treat conditions for which those drugs are known not to be effective
2. Decreased prescribing of broad-spectrum antibiotics to treat common bacterial infections.

The degree of impact in terms of prescriptions per 100 visits for each targeted outpatient infection will be compared with active education and clinical decision support versus no intervention. The study will be able to measure the value of clinical decision support with active education that will inform future efforts in disseminating outpatient antibiotic stewardship interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Clinic practices within Denver Health's Webb Center for Primary Care,
2. Clinic practices within the University of Colorado - Anschutz Campus: General Internal Medicine Clinic,
3. Clinic practices within the High Plains Network, and
4. Clinical practices within the Wilmington Health Associates System

The antibiotic prescribing patterns of primary care clinicians in these practices will be monitored over a 2 year period. Practices must be willing to assist in tracking:

1. Patient records (pediatric and adult) for conditions related to the International Classification of Diseases (ICD-9) codes associated with common infectious conditions (Upper Respiratory Infection, Acute Bronchitis, Pharyngitis, Acute Sinusitis, Otitis Media, Acute Cystitis, Cellulitis or soft tissue abscess, and Community-acquired Pneumonia) will be assessed for antibiotic prescribing,
2. 30-day events (hospitalizations,
3. Note: Emergency Department (ED) visits, or grade 3 or grade 4 abnormalities), will also be included in this study.

Exclusion Criteria:

1. Ob/Gyn related clinic visits will not be included in this study as these visits are not typically associated with high volumes of antibiotic prescribing for the infectious conditions of interest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in antibiotics prescribing behavior | December 2009 through August 2011

SECONDARY OUTCOMES:
The number and type of changes made to workflow processes when setting up or changing systems to change prescribing methods | December 2009 through August 2011

CONTACTS AND LOCATIONS:
Overall Officials: David R West, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Health and Hospitals Authority, Denver, Colorado, United States